CLINICAL TRIAL: NCT01024283
Title: Analysis of Pharmacodynamic Changes Associated With the Administration of the Heat Shock Protein 90 Inhibitor AUY922A in Patients With Advanced Solid Malignancies
Brief Title: Analysis of Pharmacodynamic Changes With AUY922A, an HSP90 Inhibitor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Dr Udai Banerji, Institute of Cancer Research
Other Study IDs: CCR3113
Record Dates: First submitted 2009-10-30; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Advanced Solid Malignancies
Keywords: Heat Shock Protein 90 Inhibitor (HSP90); Pharmacodynamic; Blood; Biopsy; Solid malignancies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The principal research objective of this additional research protocol is to support the collection, storage and use of tumour and surrogate (peripheral blood mononuclear cells - PBMNCs). The objective of this study is to perform assays to study pharmacodynamic (PD) markers that confirm target modulation.

DETAILED DESCRIPTION:
Study objectives -

1. Evaluation of HSP70, p-ERK, ERK, p-AKT and AKT in peripheral blood mononuclear cells (PBMNC). Evaluation of p-AKT and AKT will be done by commercially available Meso Scale Discovery (MSD) enzyme linked immunosorbent assay (ELISA) kits, while HSP70 will be studied using ELISA techniques developed within the Institute of Cancer Research.
2. Evaluation of HSP70, p-AKT, AKT, p-ERK, ERK, HER-2 and p-HER2 in tumour tissue. Evaluation of p-AKT, AKT, p-ERK, ERK, HER-2 and p-HER2 will be done by commercially available MSD ELISA kits, while HSP70 will be studied using ELISA techniques developed within the Institute of Cancer Research.

Study design - All patients entering the open label, phase I dose escalation and phase II expansion arms of AUY922A at the Royal Marsden Hospital will be asked to participate in this study. Patients will not have to attend additional appointments for this study and samples will be taken during visits for the planned Phase I/II clinical trial. Consent to donate samples for this research study is voluntary and patients will be asked to sign a separate consent form.

ELIGIBILITY:
Inclusion Criteria:

* All patients entering the open label phase I dose escalation and phase II expansion arms of AUY922A at the Royal Marsden Hospital will be asked to participate in this study. Patients will not have to attend additional appointments for this study and samples will be taken during visits for the planned phase I/II clinical trial.
* Consent to donate samples for this research study is voluntary and patients will be asked to sign a separate consent form.

Exclusion Criteria:

* Any patient who has not entered the open label phase I dose escalation and phase II expansion arms of AUY922A will not be asked to participate.
* Patients with advanced cancers which are not safely biopsiable will not be eligible to participate.
* Patients with known coagulation disorders.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients entering the open label phase I dose escalation and phase II expansion arms of AUY922A at the Royal Marsden Hospital will be asked to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2008-12; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
These tissues will be utilised to perform pharmacodynamic (PD) assays to demonstrate the evidence of target modulation. Together with pharmacokinetic data, scientific information from these assays will help researchers optimise drug dosing and schedule

CONTACTS AND LOCATIONS:
Overall Officials: Dr Udai Banerji, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom